CLINICAL TRIAL: NCT05315960
Title: SOcial coNNEction in Long-Term Care Home Residents
Acronym: SONNET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 146256
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Dementia
Keywords: Dementia; Long-term care; Outcome measurement; PROM; Psychometric
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative study: Consenting participants will complete a form asking about basic characteristics including age, sex, ethnicity, marital status etc. People living in long-term care and family carers will participate in an individual interview and professional staff will participate in an individual interview or focus group (between 5 and 10 participants) depending on their preference. The interview or focus group is expected to last 30-60 minutes. Sessions will be conducted in-person or online (using MS Teams), depending on preference and COVID-19-related restrictions. All sessions will be audio-recorded and transcribed.
- Cross-sectional study: Procedures:
  Consent will be obtained from residents, for those who have mental capacity to give informed consent, or from a nearest relative or caregiver as consultee, for those who lack capacity. Once consent is obtained, the LTC resident will be asked to complete a form asking about their characteristics and a questionnaire about their social connections which is expected to take approximately 15 minutes. The proxy will be asked to complete a sociodemographic form about themselves along with a number of questionnaires regarding the LTC resident's dementia severity, neuropsychiatric symptoms, activities of daily living and quality of life for comparison. Data collection for the proxy is expected to take approximately 30-60 minutes. Anticipated sample size 150 between Canada and the UK.

SUMMARY:
This study aims to develop a new measure which can accurately assess social connection for people with dementia living in long-term care homes. The Social Connection in Long-term Care home residents (SONNET) study will use interviews and focus groups with people affected by dementia and long-term care residents to establish what aspects of social connection are important for people living in care homes. These findings and a review of other studies and measures will be used to develop a new measure or measures of social connection which will then be tested in a study based in care homes in Canada and the UK.

DETAILED DESCRIPTION:
Research Question:

Can a new measure reliably and validly assess social connection for people with dementia in care homes?

Background:

Social connection, including objective and subjective constructs relating to human relationships, is a fundamental human need, but is impaired in people with dementia, particularly in those living in long-term care (LTC) settings due to cognitive impairment, complex health needs, and separation from previous social networks and community activities. Measurement instruments therefore need to be tailored to the distinct characteristics of this population and be tested in this setting, but there is no current evidence-based consensus on the best approaches to measurement.

Objectives:

1. Appraise existing measures of social connection used in LTC homes
2. Evaluate which aspects of social connection are considered important by people affected by dementia and professional staff
3. Develop a new measure informed by our appraisal of previous measures and the priorities of key stakeholders and test its preliminary psychometric properties

Methods:

A systematic review of measurement instruments assessing social connection in LTC residents, including dementia-specific measures will be conducted and measures will be appraised using COSMIN (COnsensus-based Standards for the selection of health Measurement INstruments) methodology. Focus groups and qualitative interviews will then be conducted with 50-70 people living with dementia, LTC residents, families, clinicians, care staff, and researchers in the UK and Canada to establish the important aspects of social connection and its measurement, including considerations for LTC residents with dementia and those with different stages of dementia severity. Findings from the systematic review and qualitative study will be used to inform the development of a measure or measures which will be iteratively refined during interviews. Finally, the new measure(s) will be tested for psychometric properties in 150 people with dementia living in LTC homes in the UK and Canada to establish acceptability, reliability, and validity.

ELIGIBILITY:
Qualitative study

Inclusion criteria:

* LTC residents with or without dementia: Able to provide consent for research.
* Caregivers: Visit the resident at least monthly (not including when COVID-related visitor restrictions are in place).
* Clinicians/care staff: Whose role currently includes working in LTC home or has done in past 2 years.
* Academic researchers: Have expertise in social functioning in dementia.
* All participants must be over the age of 18 years old to participate in the study.

Cross-sectional study Inclusion criteria

* LTC residents: Have a confirmed diagnosis of dementia OR Scoring ≥2 on the Noticeable Problems Checklist
* Proxy: Visit or care for the resident at least once monthly.
* All participants must be over the age of 18 years old and have adequate English language proficiency to participate in the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will purposively sample participants for diverse representation, including with respect to age, sex, gender identity, sexual orientation, socioeconomic status, race, ethnicity, and, marital status. To ensure a range of demographic characteristics and to include traditionally under-represented groups, English language proficiency for people living with dementia, LTC residents and caregivers (e.g. family, friend) is not a requirement. Interpreters will be used for those not fluent in English and arranged through the institution's interpreter services.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Resident Assessment Instrument-Minimum Data Set (RAI-MDS) Index of Social Engagement | 10 minutes
  Minimum 0, Maximum 6. Higher scores indicate a higher level of social engagement.

SECONDARY OUTCOMES:
Clinical Dementia Rating Scale | 10 minutes
  Minimum 0, Maximum 5. Higher scores indicate a more severe dementia.
Neuropsychiatric Inventory | 10 minutes
  Minimum 0, Maximum 144. Higher scores indicate a more severe neuropsychiatric symptoms.
Katz Index of Independence in activities of Daily Living | 10 minutes
  Minimum 0, Maximum 6. Higher scores indicate more independence in activities in daily living.
Dementia-specific quality of life (DEMQOL-Proxy) | 10 minutes
  Minimum 31, Maximum 124. Higher scores indicate better health-related quality of life.
Family caregiver proxy-raters only will also be asked to completed the EQ5D | 5 minutes
  Minimum 0, Maximum 1. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- University Health Network, Toronto, Ontario, Canada
- Division of Psychiatry, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chapman H, Bethell J, Dewan N, Liougas MP, Livingston G, McGilton KS, Sommerlad A. Social connection in long-term care homes: a qualitative study of barriers and facilitators. BMC Geriatr. 2024 Oct 22;24(1):857. doi: 10.1186/s12877-024-05454-8. PMID 39438797